CLINICAL TRIAL: NCT06373146
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Proof-of-Concept Study of Once-Weekly Tirzepatide Plus Mibavademab Compared With Tirzepatide Alone in Adult Participants With Obesity
Brief Title: A Study of Tirzepatide (LY3298176) Plus Mibavademab Compared With Tirzepatide Alone in Adult Participants With Obesity
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18750; I8F-MC-GPIV (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obesity
Keywords: Glucagon-like peptide-1 (GLP-1); Leptin; Incretin; Weight maintenance
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Tirzepatide (TZP) + Mibavademab (MIBA) [Group A] (Experimental): Participants will receive TZP subcutaneously (SC) and MIBA for 24 weeks. Participants in Group A will be randomized (Randomization 2) to groups C and D at week 24.
  Interventions: Drug: Tirzepatide; Drug: Mibavademab
- TZP + Mibavademab-placebo (MIBA-PBO) [Group B] (Experimental): Participants will receive TZP SC and MIBA-PBO SC for 24 weeks. Participants in Group B will be randomized (Randomization 2) to Groups E, F, G, and H at week 24.
  Interventions: Drug: Tirzepatide; Drug: Mibavademab-Placebo
- TZP + MIBA then Tirzepatide-placebo (TZP-PBO) + MIBA [Group C] (Experimental): Participants will receive TZP SC and MIBA SC for 24 weeks followed by TZP-PBO SC and MIBA SC for 24 weeks.
  Interventions: Drug: Tirzepatide; Drug: Mibavademab; Drug: Tirzepatide-Placebo
- TZP + MIBA [Group D] (Experimental): Participants will receive TZP SC + MIBA SC for 48 weeks.
  Interventions: Drug: Tirzepatide; Drug: Mibavademab
- TZP + MIBA-PBO [Group E] (Experimental): Participants will receive TZP SC + MIBA-PBO SC for 48 weeks.
  Interventions: Drug: Tirzepatide; Drug: Mibavademab-Placebo
- TZP + MIBA-PBO then TZP-PBO + MIBA [Group F] (Experimental): Participants will receive TZP SC + MIBA-PBO SC for 24 weeks followed by TZP-PBO SC + MIBA SC for 24 weeks.
  Interventions: Drug: Tirzepatide; Drug: Mibavademab; Drug: Tirzepatide-Placebo; Drug: Mibavademab-Placebo
- TZP + MIBA-PBO then TZP + MIBA [Group G] (Experimental): Participants will receive TZP SC + MIBA-PBO SC for 24 weeks followed by TZP SC + MIBA SC for 24 weeks.
  Interventions: Drug: Tirzepatide; Drug: Mibavademab; Drug: Mibavademab-Placebo
- TZP + MIBA-PBO then TZP-PBO + MIBA-PBO [Group H] (Experimental): Participants will receive TZP SC + MIBA-PBO SC for 24 weeks followed by TZP-PBO SC + MIBA-PBO SC for 24 weeks.
  Interventions: Drug: Tirzepatide; Drug: Tirzepatide-Placebo; Drug: Mibavademab-Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
Drug: Mibavademab — Administered SC
  Other Names: REGN4461
  Arms: TZP + MIBA [Group D]; TZP + MIBA then Tirzepatide-placebo (TZP-PBO) + MIBA [Group C]; TZP + MIBA-PBO then TZP + MIBA [Group G]; TZP + MIBA-PBO then TZP-PBO + MIBA [Group F]; Tirzepatide (TZP) + Mibavademab (MIBA) [Group A]
Drug: Tirzepatide-Placebo — Administered SC
  Arms: TZP + MIBA then Tirzepatide-placebo (TZP-PBO) + MIBA [Group C]; TZP + MIBA-PBO then TZP-PBO + MIBA [Group F]; TZP + MIBA-PBO then TZP-PBO + MIBA-PBO [Group H]
Drug: Mibavademab-Placebo — Administered SC
  Arms: TZP + MIBA-PBO [Group E]; TZP + MIBA-PBO then TZP + MIBA [Group G]; TZP + MIBA-PBO then TZP-PBO + MIBA [Group F]; TZP + MIBA-PBO then TZP-PBO + MIBA-PBO [Group H]; TZP + Mibavademab-placebo (MIBA-PBO) [Group B]

SUMMARY:
The main purpose of this study is to determine if combining tirzepatide with mibavademab will result in more weight loss in adult participants than tirzepatide alone. The study will last about 74 weeks and may include up to 19 visits.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≥30 kilogram/square meter (kg/m²) and ≤40 kg/m²
* Willing to learn how to self-inject study intervention (visually impaired persons who are not able to perform the injections must have the assistance of a sighted individual trained to inject the study intervention; persons with physical limitations who are not able to perform the injections must have the assistance of an individual trained to inject the study intervention)
* Male or female contraceptive use by participant should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Have a history of diabetes mellitus, including Type 1 Diabetes Mellitus (T1DM) or Type 2 Diabetes Mellitus (T2DM), history of ketoacidosis, or hyperosmolar state/coma
* Have a self-reported change (increase or decrease) in body weight >5 kilogram (kg) within 3 months prior to screening
* Have a family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia (MEN) syndrome type 2
* Have acute or chronic hepatitis
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean Percent Change from Baseline in Body Weight | Baseline, Week 48

SECONDARY OUTCOMES:
Mean Change from Baseline for Percent Change and Absolute Change in Body Weight (kg) | Baseline, Week 24
Mean Absolute Change from Baseline for Body Weight (kg) | Baseline, Week 48
Percentage of Participants Who Achieve ≥5% Body Weight Reduction | Baseline to Week 48
Percentage of Participants Who Achieve ≥10% Body Weight Reduction | Baseline to Week 48
Percentage of Participants Who Achieve ≥15% Body Weight Reduction | Baseline to Week 48
Percentage of Participants Who Achieve ≥20 Body Weight Reduction | Baseline to Week 48
Mean Percent Change from Randomization 2 for Body Weight | Week 24, Week 48
Mean Change from Randomization 2 for Body Weight (kg) | Week 24, Week 48
Mean Absolute Change from Randomization 2 for Body Weight (kg) | Week 24, Week 48
Change from Baseline to Week 24 in CoEQ Scores | Baseline, Week 24
Change from Baseline to Week 48 in CoEQ Scores | Baseline, Week 48
Change from Baseline in FCQ-T-r Scores | Baseline, Week 24
Change from Baseline in FCQ-T-r Scores | Baseline, Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (17):
- United States (17):
  - Velocity Clinical Research, Gardena, Gardena, California
  - Irvine Clinical Research, Irvine, California
  - Velocity Clinical Research, Los Angeles, Los Angeles, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Velocity Clinical Research, Santa Ana, Santa Ana, California
  - Velocity Clinical Research, Panorama City, Van Nuys, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Solaris Clinical Research, Meridian, Idaho
  - Tandem Clinical Research, Marrero, Louisiana
  - Velocity Clinical Research - New Orleans, New Orleans, Louisiana
  - Hassman Research Institute Marlton Site, Marlton, New Jersey
  - Lillestol Research, Fargo, North Dakota
  - CTI Clinical Research Center, Cincinnati, Ohio
  - South Texas Clinical Research, Corpus Christi, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - Juno Research, Houston, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Tirzepatide (LY3298176) Plus Mibavademab Compared With Tirzepatide Alone in Adult Participants With Obesity — https://trials.lilly.com/en-US/trial/477977